CLINICAL TRIAL: NCT06917105
Title: Exploratory Clinical Study on the Safety and Efficacy of CAR-T Cell Therapy in the Treatment of Relapsed/Refractory Myeloid Malignancies
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry)
Responsible Party: Principal Investigator, Jia Wei, chief physician, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202503062
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Myeloid Malignancies; CAR-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T Cells infusion（ CD33/CD123/CLL-1 CAR-T） (Experimental)
  Interventions: Drug: CD33/CD123/CLL-1 CAR-T Cells

INTERVENTIONS:
Drug: CD33/CD123/CLL-1 CAR-T Cells — Part A: Dose Escalation Phase. Follows a "3+3" dose escalation design with four predefined dose cohorts: 0.2×10⁶, 0.5×10⁶, 1×10⁶, and 2×10⁶ CAR-positive cells/kg.Anticipated enrollment: 12-24 subjects.Primary objectives: Assess safety, tolerability, and determine MTD.Dose-limiting toxicity (DLT) observation period: 28 days post-infusion.
  Part B: Dose Expansion Phase.Enrolls 21 additional subjects to receive CAR-T cell infusion at the recommended Phase 2 dose (RP2D) established in Part A.Primary objective: Further evaluate therapeutic efficacy.

SUMMARY:
This is an open-label, single-arm, exploratory clinical trial utilizing a "3+3" dose escalation followed by dose expansion to evaluate the safety, maximum tolerated dose (MTD), pharmacokinetics (PK), and preliminary efficacy of CD33/CD123/CLL-1 CAR-T cell therapy in patients with relapsed/refractory myeloid malignancies.

Part A: Dose Escalation Phase. Follows a "3+3" dose escalation design with four predefined dose cohorts: 0.2×10⁶, 0.5×10⁶, 1×10⁶, and 2×10⁶ CAR-positive cells/kg.Anticipated enrollment: 12-24 subjects.Primary objectives: Assess safety, tolerability, and determine MTD.Dose-limiting toxicity (DLT) observation period: 28 days post-infusion.

Part B: Dose Expansion Phase.Enrolls 21 additional subjects to receive CAR-T cell infusion at the recommended Phase 2 dose (RP2D) established in Part A.Primary objective: Further evaluate therapeutic efficacy.

Overall Study Objectives:Safety profile of CD33/CD123/CLL-1 CAR-T therapy.Efficacy endpoints (e.g., response rates, survival outcomes).Pharmacokinetic characterization of CAR-T cells (expansion/persistence).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: Willing and able to provide written informed consent, with commitment to comply with scheduled visits, study treatment, laboratory tests, and other trial procedures.

Age: ≥18 years, regardless of gender.

Diagnosis: Pathologically confirmed myeloid malignancy (including but not limited to AML or MDS) meeting relapsed/refractory criteria:

Relapsed Disease: Reappearance of leukemic cells in peripheral blood, bone marrow blasts >5%, or extramedullary relapse after achieving CR/CRi with ≥2 lines of salvage therapy.

Refractory Disease: Failure to achieve CR/CRi after ≥2 cycles of standard intensive chemotherapy.

Antigen Expression: Tumor cell positivity for CD33, CD123, and/or CLL-1 confirmed by immunohistochemistry (IHC) or flow cytometry.

Life Expectancy: ≥3 months from the date of informed consent signing. Hematologic Criteria: Hemoglobin ≥70 g/L (transfusion permitted).

Organ Function:

Renal: Serum creatinine ≤1.5×ULN. Cardiac: Left ventricular ejection fraction (LVEF) ≥50%. Pulmonary: Oxygen saturation >90% on room air. Hepatic: Total bilirubin ≤1.5×ULN; ALT/AST ≤2.5×ULN. Performance Status: Eastern Cooperative Oncology Group (ECOG) performance status score 0-2.

Exclusion Criteria:

* Cardiac Dysfunction: Severe cardiac insufficiency with left ventricular ejection fraction (LVEF) <50%.

Pulmonary Disease: History of severe pulmonary dysfunction (e.g., chronic respiratory failure, interstitial lung disease, or pulmonary hypertension requiring oxygen therapy).

Concurrent Malignancy: Active/progressive malignancy other than myeloid neoplasms (exceptions: adequately treated non-melanoma skin cancer or carcinoma in situ).

Uncontrolled Infection: Active severe infection requiring systemic antimicrobial therapy (antibacterial, antiviral, or antifungal) without clinical resolution.

Immune Disorders:

Severe autoimmune disease requiring immunosuppressive therapy within 6 months. Primary immunodeficiency disorders (e.g., common variable immunodeficiency, severe combined immunodeficiency).

Viral Infections:

Active hepatitis B (HBV-DNA ≥2000 IU/mL) or hepatitis C (HCV-RNA positive). HIV infection, AIDS, or untreated syphilis (confirmed by serological testing). Hypersensitivity: History of severe allergic reaction (Grade ≥3) to biological products, including antibiotics.

Transplant Complications: Allogeneic hematopoietic stem cell transplant recipients with:

Acute graft-versus-host disease (GvHD) ≥ Grade II within 3 months. Ongoing immunosuppressive therapy for GvHD within 4 weeks.

General Exclusion:

Any physical, psychiatric, or laboratory abnormality that may:

Significantly increase study risk (e.g., uncontrolled diabetes, NYHA Class III/IV heart failure).

Compromise protocol compliance or data interpretation. Investigator-determined unsuitability for trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events | Day 28

SECONDARY OUTCOMES:
Objective response rate (ORR) | At 3, 6, 9, 12, 18, and 24 months post-treatment follow up
Complete response rate (CRR) | At 3, 6, 9, 12, 18, and 24 months post-treatment follow up
Duration of response (DOR) | At 3, 6, 9, 12, 18, and 24 months post-treatment follow up
Progression free survival (PFS) | At 3, 6, 9, 12, 18, and 24 months post-treatment follow up
Overall survival (OS) | At 3, 6, 9, 12, 18, and 24 months post-treatment follow up

OTHER OUTCOMES:
Kinetics of CAR-T cells | At 3, 6, 9, 12, 18, and 24 months post-treatment follow up
  Use flow cytometry or Q-PCR to monitor the kinetics of CAR-T cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No